CLINICAL TRIAL: NCT06596174
Title: Effect of tSCS on Ankle Movement Training - Evidence From Spinal Circuitry Adaptation in Individuals With SCI
Brief Title: Effect of tSCS on Ankle Movement Training in Individuals With SCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University (Other)
Responsible Party: Principal Investigator, Ya-Ju Chang, Professor, Chang Gung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCI_001
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: SCI - Spinal Cord Injury
Keywords: post activation depression; transcutaneous spinal cord electrical stimulation (tSCS); machine-assist therapy
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1: Healthy people (Experimental): Identify optimal tSCS parameters for non-invasive spinal stimulation.
  Interventions: Procedure: Transcutaneous spinal cord stimulation (tSCS)
- Stage 2: SCI Patients (Experimental): Assess the priming effect of tSCS on spinal circuitry during machine-assisted ankle movement training.
  Interventions: Procedure: Short-term Machine-Assisted Ankle Movement Training with tSCS
- Stage 3:SCI Patients (Experimental): Long-term clinical effects of combined tSCS and ankle movement training
  Interventions: Procedure: Long-term Effects of Machine-Assisted Ankle Movement Training with tSCS
- Stage 3:SCI Patients(Control) (No Intervention): Control Group

INTERVENTIONS:
Procedure: Transcutaneous spinal cord stimulation (tSCS) — The subjects will undergo 20 minutes transcutaneous spinal cord stimulation (tSCS).
  Arms: Stage 1: Healthy people
Procedure: Short-term Machine-Assisted Ankle Movement Training with tSCS — The subjects will undergo 30 minutes of machine-assisted ankle movement training combined with transcutaneous spinal cord stimulation (tSCS) at a time
  Arms: Stage 2: SCI Patients
Procedure: Long-term Effects of Machine-Assisted Ankle Movement Training with tSCS — The subjects will undergo machine-assisted ankle movement training combined with transcutaneous spinal cord stimulation (tSCS).
  Each session will last for 30 minutes, conducted three times per week, over a period of four weeks.
  Arms: Stage 3:SCI Patients

SUMMARY:
This clinical trial explores the effectiveness of transcutaneous spinal cord stimulation (tSCS), a non-invasive technique, in facilitating spinal circuitry adaptation in individuals with spinal cord injury (SCI). While epidural spinal cord stimulation (eSCS) has shown functional benefits, its application is limited by the side effects associated with implanted electrodes. tSCS, which shares a similar mechanism but does not require surgery, has yet to be extensively studied in large human trials.

The study aims to:

Determine optimal tSCS parameters for non-invasive spinal stimulation. Investigate the priming effect of tSCS on spinal circuitry during machine-assisted ankle movement training.

Examine the long-term clinical outcomes of combining tSCS with ankle movement training in individuals with incomplete SCI.

The trial will include both healthy participants and individuals with complete and incomplete SCI, using the soleus post-activation depression (PAD) model to evaluate spinal circuitry adaptation. The results will provide insights into spinal re-adaptation and potentially introduce a novel, non-invasive approach for SCI rehabilitation.

ELIGIBILITY:
Health subjects:

Exclusion Criteria:

1. Musculoskeletal injuries on legs.
2. Osteoporosis.

SCI subjects:

Inclusion Criteria

1. Participants with chronic spinal cord injury, with injury duration greater than one year.

Exclusion Criteria

1. Current musculoskeletal or joint injuries in the lower limbs.
2. History of central or peripheral neuromuscular diseases.
3. Presence of a pacemaker.
4. Current use of antispastic or antidepressant medications.
5. Current venous thromboembolism or osteoporosis.
6. Impairment of the soleus H-reflex arc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Latency and amplitude of the H-reflex | Baseline, 4 weeks
  The H-reflex will be elicited through electrical stimulation of the tibial nerve (or sciatic nerve) using electromyography (EMG) to record the resulting muscle response.
Latency, amplitude, and duration of the M-wave | Baseline, 4 weeks
  The M-wave will be elicited by direct electrical stimulation of the motor nerve (e.g., tibial nerve) and recorded using electromyography (EMG) from the target muscle (e.g., soleus muscle).
Level of Post-Activation Depression (PAD) of the H-reflex | Baseline, 4 weeks
  The H-reflex will be elicited by electrical stimulation of the tibial nerve (or other motor nerves), and PAD will be assessed by measuring the reduction in H-reflex amplitude following a series of repetitive stimuli. The amplitude of the H-reflex after repeated stimulation will be compared to the baseline single stimulus.
Latency and amplitude of the Posterior Root Muscle (PRM) reflex | Baseline, 4 weeks
  The PRM reflex will be elicited by stimulating the posterior roots of the spinal cord (typically via electrical stimulation of the dorsal roots), and the resulting muscle activity will be recorded using electromyography (EMG)
Muscle spasticity levels as assessed by the Modified Ashworth Scale (MAS). | Baseline, 4 weeks
  Muscle spasticity will be evaluated using the MAS, which grades the resistance encountered during passive movement of the affected limb (e.g., arm or leg). The scale ranges from 0 (no increase in muscle tone) to 4 (affected part rigid in flexion or extension).
Muscle Tone (Frequency, Hz) | Baseline, 4 weeks
  This parameter measures the natural oscillation frequency of the muscle in response. It reflects the muscle's state of tension or readiness.
Elasticity (Dynamic Stiffness, N/m) | Baseline, 4 weeks
  Elasticity, measured in Newtons per meter, reflects the muscle's ability to return to its original shape after being deformed by the impulse
Stiffness (Decay, ms) | Baseline, 4 weeks
  This parameter quantifies the rate at which the muscle returns to its initial state after the impulse, indicating the muscle's stiffness
Mechanical Stress (Creep, s) and Relaxation (S) | Baseline, 4 weeks
  These parameters measure the time it takes for muscle tissue to adapt to a sustained force (creep) and the time it takes for the muscle to return to a relaxed state after removing the force (relaxation).

SECONDARY OUTCOMES:
Foot pressure distribution and peak pressure. | Measured continuously during CPM
  Foot pressure will be measured using pressure sensors during ankle movement
The score of 10-meter walking test (10MWT) | Baseline, 4 weeks.
  To measure walking speed over a short distance as a quantitative index of walking ability.
Ankle Joint Range of Motion (ROM) | Baseline, 4 weeks
  These movements measure the ability to move the foot up towards the shin (dorsiflexion) and down away from the body (plantarflexion). Typical instruments used include a universal goniometer or an inclinometer. The patient is typically seated or lying down with the knee extended for accurate measurement.
Knee Joint ROM | Baseline, 4 weeks
  These are the primary movements of the knee, involving bending (flexion) and straightening (extension) of the leg. Measurements are taken with the patient seated or lying down. A goniometer is placed on the lateral aspect of the knee to record the angle of maximum bend and extension.
Overall the Patient Reported Impact of Spasticity Measure(PRISM) Score | Baseline, 4 weeks
  An aggregated score derived from all the individual items within the questionnaire, providing a comprehensive measure of the impact of spasticity on the patient's quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan